CLINICAL TRIAL: NCT05550896
Title: Platelet Adhesion in the Pathobiology of Aortic Stenosis
Status: Recruiting | Type: Observational
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Jonathan Lindner, MD, Professor of Medicine, Vice Chief for Research, Cardiovascular Division, University of Virginia
Other Study IDs: HSR220332
Record Dates: First submitted 2022-09-19; First posted 2022-09-22 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mild to moderate AS: Patients with mild to moderate AS by echocardiography
  Interventions: Diagnostic Test: Echocardiogaphy
- Controls: Age and sex match controls with no AS by echocardiography
  Interventions: Diagnostic Test: Echocardiogaphy

INTERVENTIONS:
Diagnostic Test: Echocardiogaphy — Assessment of high velocity low amplitude signals on Doppler echocardiography

SUMMARY:
Aortic stenosis (AS) is a serious and common condition that affects 2-3% of the population >65 years of age in Western countries. It is also responsible for extraordinarily high healthcare expenditures, estimated to be over $6 billion annually,2 in part because the primary treatment for severe AS is aortic valve replacement (AVR) which is resource-intensive. Valve abnormalities are frequently recognized before AS becomes severe, or before there is need for guideline-directed procedural intervention, thereby providing an opportunity for pharmacologic intervention to slow disease progression. Yet, all attempts to prevent AS progression in those with degenerative non-congenital forms of disease have failed. The only non-procedural intervention that benefits patients with moderate or greater AS is the aggressive treatment of hypertension, which reduces net left ventricular (LV) afterload (valvulo-arterial impedance [Zva]) and can slow secondary LV remodeling. The overall goal of this proposal is to integrate advanced imaging and vascular biology to study how von Willebrand factor (VWF) and platelet adhesion promote AS progression through many parallel pathways, thereby representing a potential therapeutic target. We are hypothesizing that blood markers of abnormal VWF proteolysis and platelet-derived factors, and abnormal valve shear patterns which can be detected by advanced analysis of spectral Doppler on echocardiography are predictors for progressive AS.

ELIGIBILITY:
Inclusion Criteria For AS group

* Age >25 years of age
* Mild or moderate calcific, non-congenital aortic stenosis by echocardiography within the prior 3 months defined as:

  * aortic valve area 1.0 cm2 - 1.9 cm2 and either
  * peak velocity of >2.5 m/s and <4.0 m/s with normal or mildly reduced stroke volume index (>25 ml/m2), or
  * VTI ratio (LVOT:AoV) of <0.5 and >0.25 with abnormal stroke volume (<35 ml/m2 or >60 ml/m2).
* Age and sex-matched control subjects undergoing echocardiography with no aortic stenosis, and no more than mild severity disease of other valves.

Inclusion criteria for Control Group

Exclusion Criteria:

-

Min Age: 25 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: * Age-matched to the Aortic Valve Disease group
  * Referred for echocardiography for a clinical indication
  * Absence of valve disease
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2023-01-03 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Evidence for High Shear Patterns on Echocardiography | 4 years
  Low-amplitude high velocity signals on spectral Doppler

SECONDARY OUTCOMES:
Plasma markers of VWF | 4 years
  Plasma markers including VWF antigen, oxidation, cleavage; and ADAMTS13 activity

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ozawa K, Muller MA, Varlamov O, Hagen MW, Packwood W, Morgan TK, Xie A, Lopez CS, Chung D, Chen J, Lopez JA, Lindner JR. Reduced Proteolytic Cleavage of von Willebrand Factor Leads to Aortic Valve Stenosis and Load-Dependent Ventricular Remodeling. JACC Basic Transl Sci. 2022 Jun 29;7(7):642-655. doi: 10.1016/j.jacbts.2022.02.021. eCollection 2022 Jul. PMID 35958695